CLINICAL TRIAL: NCT01690949
Title: Single-blind Evaluation of the Effect of PUR118 on Ozone Induced Airway Inflammation in Healthy Normal Volunteers
Brief Title: Evaluation of the Effect of PUR118 on Ozone Induced Airway Inflammation in Healthy Normal Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pulmatrix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 601-0005
Record Dates: First submitted 2012-09-12; First posted 2012-09-24 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: inflammation; COPD; respiratory disease; healthy volunteers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation; Respiration Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- PUR118 low dose (Experimental)
  Interventions: Drug: PUR118
- PUR118 mid dose (Experimental)
  Interventions: Drug: PUR118
- PUR118 high dose (Experimental)
  Interventions: Drug: PUR118

INTERVENTIONS:
Drug: PUR118 — inhaled PUR118, BID

SUMMARY:
This trial in healthy subjects will assess PUR118's effect on attenuating ozone induced airway inflammation. This trial will establish the tolerability of PUR118 in healthy normal volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non pregnant, non lactating healthy females age 18-50 years;
* Must be able to produce acceptable sputum sample by induction;
* Must respond to ozone inhalation with a > 10% increase in the absolute percentage of sputum neutrophils and the total neutrophils (neutrophils/gram sputum) must increase by at least 50% from the sputum neutrophil count at screening;
* Volunteer is a non-smoker or ex-smoker of at least 12 months' duration prior to screening with a history of less than 1 pack per year.

Exclusion Criteria:

* Volunteers receiving chronic medication other than oral contraceptives;
* Screening forced expiratory volume FEV1 is < 80% of the predicted value for their age, gender, height and race and/or their FEV1/FVC ration is below 70%;
* Volunteers with significant occupational exposure to respiratory irritants or toxins
* Upper respiratory tract infection within 30 days of the first study day, or lower respiratory tract infection within the last 3 months;
* Volunteers taking any medication that may affect the respiratory tract within 30 days of the first study day;
* Volunteers with a history of asthma

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sputum cell counts and inflammatory markers | 6 hours post-initiation of ozone challenge
Change from baseline in white blood cell and inflammatory biomarker counts in blood | 7 and 24 hours post-initiation of ozone challenge

SECONDARY OUTCOMES:
Change from baseline in pulmonary function | all post-dose timepoints up to 24 hours post-initiation of ozone challenge
Changes in clinical signs and symptoms from physical examination at baseline | Subjects will be followed for an expected average of 12 weeks
Changes in clinical safety laboratory tests from baseline | Subjects will be followed for an expected average of 12 weeks
Changes in vital signs from baseline | Subjects will be followed for an expected average of 12 weeks
Changes in ECG from baseline | Subjects will be followed for an expected average of 12 weeks
Number of subjects with adverse events | Subjects will be followed for an expected average of 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Hanrahan, MD, Study Director — Pulmatrix Inc.
Locations (1):
- Fraunhofer Institut fur Toxicologie und Experimentelle Medicine (ITEM), Hanover, Germany

REFERENCES:
- [Derived] Holz O, Biller H, Mueller M, Kane K, Rosano M, Hanrahan J, Hava DL, Hohlfeld JM. Efficacy and safety of inhaled calcium lactate PUR118 in the ozone challenge model--a clinical trial. BMC Pharmacol Toxicol. 2015 Aug 12;16:21. doi: 10.1186/s40360-015-0021-1. PMID 26265479